CLINICAL TRIAL: NCT03788096
Title: Peer Support for Post Intensive Care Syndrome Self-Management (PS-PICS)
Brief Title: Peer Support for Post Intensive Care Syndrome Self-Management
Acronym: PS-PICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Valerie Danesh, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-08-0097
Record Dates: First submitted 2018-11-20; First posted 2018-12-27 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Critical Illness; Sepsis; Shock, Septic; Shock; Respiratory Failure; Respiratory Distress Syndrome, Adult; Shock, Hypovolemic; Chronic Disease
Keywords: Post-Intensive Care Syndrome (PICS); Chronic Critical Illness
MeSH Terms: conditions — Critical Illness; Sepsis; Shock, Septic; Shock; Respiratory Insufficiency; Respiratory Distress Syndrome; Chronic Disease; postintensive care syndrome | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A prospective, 2-arm, single-blind, randomized controlled clinical feasibility trial design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PS-PICS Peer Support Intervention (Experimental): ICU mentors will be responsible for providing support to survivor participants randomized to the PS-PICS peer support intervention. Mentors will be trained in motivational interviewing techniques to engage mentees in goal setting and emotional management that is not readily accessible as part of discharge planning.
  Interventions: Behavioral: Peer Support with Motivational Interviewing
- Usual Care Group (Placebo Comparator): A control intervention will be used to provide comparison data consistent with usual care (absence of structured peer support telephone intervention) to evaluate the impact of the PS-PICS peer support intervention.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: Peer Support with Motivational Interviewing — Mentors will trained in motivational interviewing and will conduct weekly telephone calls with participants randomized to the PS-PICS peer support intervention arm.
  Arms: PS-PICS Peer Support Intervention
Behavioral: Usual Care Group — Usual care.
  Arms: Usual Care Group

SUMMARY:
A prospective, 2-arm, single-blind, randomized controlled clinical feasibility trial design is planned. Forty CCI survivors will be randomized (1:1) to either the PS-PICS (peer support) intervention or usual care (control) group.

DETAILED DESCRIPTION:
Randomized participants will complete 4 study assessments: 1) baseline data at hospital discharge; 2) baseline data post-hospital discharge and before the start of the weekly peer support intervention; 3) post-intervention at the conclusion of the 90-day weekly peer support intervention; and 4) follow-up at 6-months post-hospital discharge. The weekly peer support intervention will be delivered by a small pool of critical illness survivor peers (mentors) recruited from the study site from previous research. Peer support mentors will be trained in peer support and MI, and will deliver 3 months of weekly MI interventions (phone-based) to CCI survivors randomized to the intervention group. Participants randomized to the usual care group will not receive the weekly peer support/MI intervention but will receive the usual discharge planning services currently provided at hospital discharge. Participants in both groups will be contacted by the research team for 4 telephone-based assessments. The design will allow us to test the feasibility and potential impact of the PS-PICS intervention on social relationship measures, depression and self-management. Data collection and analyses are guided by the Individual and Family Self-Management Theory. The Individual and Family Self-Management Theory illustrates the interaction of the process of self-management with risk and protective factors, and short-term and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age18 years or older
* ICU length of stay 8 days or longer
* expected to survive hospitalization with a discharge destination to home within 28 days of hospital discharge
* diagnosed with 2 or more chronic conditions.

Exclusion Criteria:

* death prior to hospital discharge
* enrollment in Hospice services at the time of hospital discharge
* non-communicative
* no access to telephone
* incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-10-27 (Estimated); Study Completion 2021-01-27 (Estimated)

PRIMARY OUTCOMES:
Social Network Index | 3 months post-intervention
  Social Network Index (SNI) to measure social relationships. The scale range is 0-12. The total score will be reported. The maximum total score is 12. Higher values represent a broader diversity of social networks and are classified as a better outcome.

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D) | 1-week Post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D) to measure self-reported symptoms of depression The scale range is 0-60. The total score will be reported. The maximum total score is 60. Higher values represent self-reported symptoms of depression. Higher values represent a worse outcome.
Center for Epidemiologic Studies Depression Scale (CES-D) | 3 months post-intervention
  Center for Epidemiologic Studies Depression Scale (CES-D) to measure self-reported symptoms of depression The scale range is 0-60. The total score will be reported. The maximum total score is 60. Higher values represent self-reported symptoms of depression. Higher values represent a worse outcome.
Social Network Index | 1-week Post-intervention
  Social Network Index (SNI) to measure social relationships. The scale range is 0-12. The total score will be reported. The maximum total score is 12. Higher values represent a broader diversity of social networks and are classified as a better outcome.
Patient Activation Measure | 1-week Post-intervention
  Patient Activation Measure (PAM) Survey to measure self-reported active behavior in the self-management of chronic illness.
  The scale range is 0-100. The total score will be reported. The maximum total score is 100. Higher values represent high levels of activation in self-management. Higher values represent a better outcome.
Patient Activation Measure | 3 months post-intervention
  Patient Activation Measure (PAM) Survey to measure self-reported active behavior in the self-management of chronic illness.
  The scale range is 0-100. The total score will be reported. The maximum total score is 100. Higher values represent high levels of activation in self-management. Higher values represent a better outcome.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale | 1-week Post-intervention
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale The scale range is 0-65. The total score will be reported. For each scale range provided, specify which values are considered to be a better or worse outcome (e.g., Do higher values represent a better or worse outcome?).
  The maximum total score is 65. Higher values represent higher levels of fatigue.
Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale | 3 months post-intervention
  The Measure includes a scale. Please provide the following scale information:
  Specify the full (unabbreviated) scale name and construct (i.e., indicate what the scale measures if not clear from name).
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale Include all scale ranges (i.e., minimum and maximum scores) required to interpret any values. For example, if the *total* score is reported, the *total* range should be provided. If *subscale* scores are reported, the range for each *subscale* should be provided.
  The scale range is 0-65. The total score will be reported. For each scale range provided, specify which values are considered to be a better or worse outcome (e.g., Do higher values represent a better or worse outcome?).
  The maximum total score is 65. Higher values represent higher levels of fatigue.
  If subscales are combined to compute a total score, consider indicating how subscales are combined (summed, averaged, etc.).
  N/A
Short Form-36 (SF-36) | 1-week Post-intervention
  Short Form-36 (SF-36) or 36-Item Short Form Health Survey Instrument The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100.
  Lower scores = more disability, higher scores = less disability Sections: ∙ Vitality ∙ Physical functioning ∙ Bodily pain ∙ General health perceptions ∙ Physical role functi
Short Form-36 (SF-36) | 3 months post-intervention
  Short Form-36 (SF-36) or 36-Item Short Form Health Survey Instrument The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100.
  Lower scores = more disability, higher scores = less disability Sections: ∙ Vitality ∙ Physical functioning ∙ Bodily pain ∙ General health perceptions ∙ Physical role functi

OTHER OUTCOMES:
Health services utilization | 1-week Post-intervention
  Utilization of health services
Health services utilization | 3 months post intervention
  Utilization of health services

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Health, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided